CLINICAL TRIAL: NCT05407779
Title: An Open-Label, Non-controlled Study of the Pharmacodynamics, Pharmacokinetics, Safety, and Immunogenicity of Single Escalating Doses of BCD-180 (JSC BIOCAD, Russia) in Healthy Volunteers
Brief Title: Study of the Pharmacodynamics, Pharmacokinetics, Safety, and Immunogenicity of Single Escalating Doses of BCD-180 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BCD-180-1
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Stage 1. The first cohort will include one subject ("sentinel volunteer") who will receive BCD-180 at a dose 1. Starting from the 2nd cohort, the study will have a classic "3 + 3" design.
  Subjects will be monitored for 14 days following drug administration to assess the presence of dose limiting toxicity (DLT). In the absence of DLT, another cohort with a higher dose level will be formed.
  After all subjects have completed the main study period (Days 1-57), the safe dose range of BCD-180 will be determined based on assessed PD, PK, safety and immunogenicity endpoints.
  Further follow-up of the subjects included in stage 1 will continue up to a year.
  Stage 2. Two cohorts of healthy Asian volunteers (Cohorts 8 and 9) will be included. Subjects will receive a single infusion of BCD-180 at selected doses planned for further clinical development based on the results of the main period of stage 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): The Cohort 1 include one subject ("sentinel volunteer") to receive BCD-180 at a dose 1
  Interventions: Biological: BCD-180, dose 1
- Cohort 2 (Experimental): The Cohort 2 include 3 subjects to receive BCD-180 at a dose 2
  Interventions: Biological: BCD-180, dose 2
- Cohort 3 (Experimental): The Cohort 3 include 3 subjects to receive BCD-180 at a dose 3
  Interventions: Biological: BCD-180, dose 3
- Cohort 4 (Experimental): The Cohort 4 include 3 subjects to receive BCD-180 at a dose 4
  Interventions: Biological: BCD-180, dose 4
- Cohort 5 (Experimental): The Cohort 5 include 3 subjects to receive BCD-180 at a dose 5
  Interventions: Biological: BCD-180, dose 5
- Cohort 6 (Experimental): The Cohort 6 include 3 subjects to receive BCD-180 at a dose 6
  Interventions: Biological: BCD-180, dose 6
- Cohort 7 (Experimental): The Cohort 7 include 3 subjects to receive BCD-180 at a dose 7
  Interventions: Biological: BCD-180, dose 7
- Cohort 8 (Experimental): The Cohort 8 include 3 subjects to receive BCD-180 at one of two selected for the further development doses
  Interventions: Biological: BCD-180, dose 6
- Cohort 9 (Experimental): The Cohort 9 include 3 subjects to receive BCD-180 at one of two selected for the further development doses
  Interventions: Biological: BCD-180, dose 7

INTERVENTIONS:
Biological: BCD-180, dose 1 — anti-TRBV9 monoclonal antibody single infusion at dose 1
  Arms: Cohort 1
Biological: BCD-180, dose 2 — anti-TRBV9 monoclonal antibody, single infusion at dose 2
  Arms: Cohort 2
Biological: BCD-180, dose 3 — anti-TRBV9 monoclonal antibody, single infusion at dose 3
  Arms: Cohort 3
Biological: BCD-180, dose 4 — anti-TRBV9 monoclonal antibody, single infusion at dose 4
  Arms: Cohort 4
Biological: BCD-180, dose 5 — anti-TRBV9 monoclonal antibody, single infusion at dose 5
  Arms: Cohort 5
Biological: BCD-180, dose 6 — anti-TRBV9 monoclonal antibody, single infusion at dose 6
  Arms: Cohort 6; Cohort 8
Biological: BCD-180, dose 7 — anti-TRBV9 monoclonal antibody, single infusion at dose 7
  Arms: Cohort 7; Cohort 9

SUMMARY:
The aim of the study is to investigate the pharmacodynamics, pharmacokinetics, safety, and immunogenicity of BCD-180 after a single intravenous administration in escalating doses to healthy volunteers.

DETAILED DESCRIPTION:
The study will be carried out in 2 stages. Stage 1 involves administration of escalating doses of study drug (BCD-180) in 7 cohorts of healthy subjects. The first cohort will include one subject ("sentinel volunteer"). Each of the subsequent cohorts will include 3 subjects, each of whom will receive a preset cohort dose of BCD-180 as a single intravenous infusion. Stage 2: additionally two cohorts of healthy Asian volunteers (Cohorts 8 and 9) will be included: subjects will receive a single infusion of BCD-180 at selected doses (planned for further clinical development) based on the results of the main period of Stage 1.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent form (ICF) for participation in the study.
2. Men aged 18 to 45 inclusive at the time of ICF signing.
3. For stage 2: Asian race.
4. The ability of the subject to follow the Protocol procedures, according to the investigator.
5. A diagnosis of "health" established using standard clinical, laboratory tests and investigations carried out at screening, according to the investigator, as well as medical history data (no acute or chronic respiratory, gastrointestinal, cardiovascular, nervous system diseases, hepatic or renal impairment).
6. Hemodynamic parameters within normal limits: systolic blood pressure (SBP) within 100-130 mm Hg, diastolic blood pressure (DBP) within 60-90 mm Hg, pulse rate within 60-90 bpm.
7. Willingness of subjects and their female sexual partners of childbearing potential to use reliable contraception from the ICF signing throughout the main period of the study and during Day 57 of the main period of the study. This requirement does not apply to subjects who have had surgical sterilization. Reliable methods of contraception involve the use of one barrier method in combination with one of the following in the female partner: spermicides, intrauterine device/oral contraceptives.
8. Willingness to refrain from participating in any other clinical trials, starting from the ICF signing, throughout the main study period and during Day 57 of the main study period, and in other clinical trials involving the administration of any drugs that affect the human immune system, including other monoclonal antibody products with immunosuppressive action, during the current study, i.e., until the end of participation in it.

Exclusion Criteria:

1. Any medical or social condition that, in the opinion of the investigator, precludes participation in this study.
2. Any confirmed or suspected immunosuppressive or immunodeficient condition.
3. Any acute infectious or non-infectious disease, including convalescence, less than 4 weeks from clinical recovery, as well as during the screening.
4. A diagnosis of infectious mononucleosis (either documented or reported by the subject) made within 2 months prior to the ICF signing or during the screening.
5. BCG (Bacillus Calmette-Guérin vaccine) vaccination (within 12 weeks), administration of live vaccines (within 8 weeks) or any other vaccines (within 4 weeks) before signing the ICF or during the screening.
6. Medical history of allergic reactions and evidence of other significant adverse reactions after administration of any medicinal products.
7. Hypersensitivity to any of the BCD-180 ingredients or premedication drugs.
8. Body mass index (BMI) outside of the normal range (18.0-30.0 kg/m2).
9. Results of standard laboratory and imaging tests that fall beyond the reference intervals adopted at the study center.
10. Positive screening tests for HIV infection, hepatitis B and C, syphilis, tuberculosis.
11. Positive urine test for psychotropic, narcotic, psychoactive drugs or saliva alcohol test at screening.
12. Impossibility of venipuncture to collect blood samples (for example, due to skin disease at venipuncture sites).
13. Long-term (more than 14 days) use of drugs that have a pronounced effect on hemodynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, etc.) less than 30 days before the ICF signing; prior use of drugs that affect the immune system, including other monoclonal antibody products, with immunosuppressive action.
14. Regular oral or parenteral administration of any medicinal products, including over-the-counter drugs, vitamins and dietary supplements, less than 14 days before the ICF signing.
15. Smoking more than 10 cigarettes a day.
16. Consumption of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ L of beer, 200 mL of wine or 20 mL of spirits) or a history of alcoholism, drug addiction or drug abuse.
17. Surgical interventions performed less than 90 days before the ICF signing.
18. Donation of 450 mL or more of blood or plasma within 60 days prior to the ICF signing.
19. Participation in any clinical studies of medicinal products less than 90 days prior to the ICF signing; previous participation in this study in case of administration of the investigational product .
20. For stage 2: a history of coronavirus infection (positive polymerase chain reaction (PCR) test for SARC-CoV2-RNA) within 8 weeks prior to the ICF signing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with adverse reactions | 361 days after the study drug administration for stage 1
Proportion of subjects with adverse reactions | 57 days after the study drug administration for stage 2

OTHER OUTCOMES:
Proportion of subjects with serious adverse reactions | 361 days after the study drug administration for stage 1
Proportion of subjects with serious adverse reactions | 57 days after the study drug administration for stage 2
Proportion of subjects with adverse reactions of grade 3 or higher according to CTCAE 5.0 | 361 days after the study drug administration for stage 1
Proportion of subjects with adverse reactions of grade 3 or higher according to CTCAE 5.0 | 361 days after the study drug administration for stage 2
Proportion of subjects who prematurely withdrew from the study due to adverse reactions | 361 days after the study drug administration fo stage 1
Proportion of subjects who prematurely withdrew from the study due to adverse reactions | 57 days after the study drug administration fo stage 2
Proportion of Binding antibodies (BAb) and neutrolizing antibodies (NAb) positive subjects | 361 days after the study drug administration
Proportion of Binding antibodies (BAb) and neutrolizing antibodies (NAb) positive subjects | 361 days after the study drug administration fo stage 1
Titer of BAb and/or NAb | 361 days after the study drug administration for stage 1
Titer of BAb and/or NAb antibodies | 57 days after the study drug administration for stage 2
AUC 0-1344 | day 57
  Area under the concentration-time curve from administration to Day 57 (1344 hours)
AUC0-2016 | day 85
  Area under the concentration-time curve from administration to Day 85 (2016 hours) (for stage 1)

CONTACTS AND LOCATIONS:
Locations (1):
- X7 Clinical Research, Saint Petersburg, Russia